CLINICAL TRIAL: NCT04736550
Title: Enhancing Exercise and Psychotherapy to Treat Pain and Addiction in Adults With an Opioid Use Disorder (EXPO): A Randomized Pilot Trial
Brief Title: Enhancing Exercise and Psychotherapy to Treat Pain and Addiction in Opioid Use Disorders ("EXPO" Pilot Trial)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: University of Colorado, Denver (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Nora Nock, Associate Professor, Case Western Reserve University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY20201427; R61AT010806 (NIH)
Record Dates: First submitted 2021-01-27; First posted 2021-02-03 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Opioid-use Disorder; Pain
Keywords: exercise; psychotherapy; residential drug treatment; OUD; chronic pain
MeSH Terms: conditions — Opioid-Related Disorders; Pain; Motor Activity; Chronic Pain | interventions — Exercise; Psychotherapy

STUDY DESIGN:
Intervention Model Description: In the pilot trial (R61 Phase), the investigators will use a multi-phase optimization trial (MOST) approach to help identify which components of the exercise and psychotherapy for pain treatment program are viable and worth retaining in the planned fully powered trial (R33 Phase). In the R61 Phase/Pilot Trial, the investigators will have two intervention components: 1) exercise with 3 levels ('assisted', voluntary, none/treatment as usual (TAU); and, 2) psychotherapy for pain (I-STOP) with 2 levels (Yes/I-STOP, No/TAU). All participants will receive also receive the treatment as usual at their residential drug treatment program and any medication assisted treatment (MAT). This corresponds to a 2^1 x 3 1 full factorial with six experimental conditions.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Assisted Exercise and I-STOP (Experimental): Participant will receive Assisted Exercise (stationary cycling) and psychotherapy for pain (I-STOP). Exercise (supervised) will be offered 3 days/week. I-STOP will be offered 1 day/week.
  Interventions: Behavioral: Exercise; Behavioral: Psychotherapy for Pain (I-STOP)
- Voluntary Exercise and I-STOP (Experimental): Participant will receive Voluntary Rate Exercise (stationary cycling) and psychotherapy for pain (I-STOP). Exercise (supervised) will be offered 3 days/week. I-STOP will be offered 1 day/week.
  Interventions: Behavioral: Exercise; Behavioral: Psychotherapy for Pain (I-STOP)
- No Exercise (TAU) and I-STOP (Experimental): Participant will receive psychotherapy for pain (I-STOP). I-STOP will be offered 1 day/week.
  Interventions: Behavioral: Psychotherapy for Pain (I-STOP)
- Assisted Exercise and No I-STOP (TAU) (Experimental): Participant will receive Assisted Exercise (stationary cycling). Exercise (supervised) will be offered 3 days/week.
  Interventions: Behavioral: Exercise
- Voluntary Exercise and No I-STOP (TAU) (Experimental): Participant will receive Voluntary Rate Exercise (stationary cycling). Exercise (supervised) will be offered 3 days/week.
  Interventions: Behavioral: Exercise
- No Exercise (TAU) and No I-STOP (TAU) (No Intervention): Participant will receive their usual behavioral treatment offered at the residential drug treatment center and their medicated assisted treatment (MAT) as applicable.

INTERVENTIONS:
Behavioral: Exercise — Participants who are randomized to exercise will be perform exercise on stationary bikes. Participants randomized to "Voluntary Exercise" will exercise on a standard stationary bike where they will pedal at their voluntary rates. Participants randomized to "Assisted Exercise" will exercise on a special bike that assists them to pedal faster than they do voluntarily on their own ("assisted (exercise) bike").
  Arms: Assisted Exercise and I-STOP; Assisted Exercise and No I-STOP (TAU); Voluntary Exercise and I-STOP; Voluntary Exercise and No I-STOP (TAU)
Behavioral: Psychotherapy for Pain (I-STOP) — Participants who are randomized to receive I-STOP will receive the "Self-regulation Treatment for Opioid addiction and Pain" (STOP) program modified for inpatients/residential drug treatment (I-STOP). I-STOP uses empirically validated pain psychotherapy approaches targeted to patients with an OUD using psycho-physiological self-regulation components and biofeedback with "Bio-dots".
  Arms: Assisted Exercise and I-STOP; No Exercise (TAU) and I-STOP; Voluntary Exercise and I-STOP

SUMMARY:
The purpose of this pilot trial is to determine the feasibility of integrating exercise and psychotherapy that is specifically targeted to reducing and managing pain into residential drug treatment programs. The investigators will evaluate the feasibility (adherence) of integrating 'assisted' rate cycling, voluntary rate cycling and psychotherapy for pain (I-STOP) in participants with an opioid use disorder (OUD) and pain enrolled in residential drug treatment programs. The investigators will also explore the potential effects of 'assisted' rate cycling, voluntary rate cycling and I-STOP on pain, cravings, depression, anxiety, weight and sleep.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* Must be enrolled in a Residential Drug Treatment Program at a collaborating drug treatment center
* Must be diagnosed with an Opioid Use Disorder (OUD; ICD-10 F11.20) or a Poly-substance Drug Use that includes an opioid component (ICD-10,F19.xx) and self-reported pain or a pain condition describing a non-cancer related chronic pain disorder
* Must be approved to exercise in the study by the drug treatment center Medical Director, physician or other relevant clinical staff or primary care physician (PCP)

Exclusion Criteria:

* Any substantive contraindications to exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence (% of sessions attended) | through study completion, an average of 8 weeks
  Percentage of exercise and psychotherapy sessions attended

SECONDARY OUTCOMES:
Change in pain | baseline/pre-intervention and immediately after the intervention
  The investigators will evaluate potential changes in pain using a cold pressor pain task. Pain sensitivity is the time spent in a cold water bath until the first report of pain and pain tolerance is the total time in the cold water bath.
Change in weight | baseline/pre-intervention and immediately after the intervention
  The investigators will evaluate potential changes in weight (lbs).
Change in depression | baseline/pre-intervention and immediately after the intervention
  The investigators will evaluate potential changes in depression using self-report, standardized questionnaire (Depression sub-scale in Hospital Anxiety and Depression Scale, HADS). Total Score range: 0-21; Higher scores indicate higher levels of depression.
The investigators will evaluate potential changes in drug cravings using self-report visual analog scale (VAS) | baseline/pre-intervention and immediately after the intervention
  Higher scores indicate higher levels of cravings.
Change in cravings assessed by standardized questionnaire (Desires for Drug Questionnaire) | baseline/pre-intervention and immediately after the intervention
  Higher scores indicate higher levels of cravings.
Change in sleep | baseline/pre-intervention and immediately after the intervention
  The investigators will evaluate potential changes in sleep using self-report, standardized questionnaire (Pittsburgh Sleep Quality Index, PSQI). Total Score range: 0-21; Higher scores indicate poorer sleep quality.
Change in Anxiety | baseline/pre-intervention and immediately after the intervention
  The investigators will evaluate potential changes in depression using self-report, standardized questionnaire (Anxiety sub-scale in Hospital Anxiety and Depression Scale, HADS). Total Score range: 0-21; Higher scores indicate higher levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Nora L Nock, PhD, Principal Investigator — Case Western Reserve University
Locations (2):
- United States (2):
  - University of Colorado at Denver, Denver, Colorado
  - Case Western Reserve University, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No